CLINICAL TRIAL: NCT02245061
Title: Cortical Excitability Assessment of Pharmacoresistant Focal Epilepsy Using Direct Electrical Stimulation During Stereo-electroencephalography
Brief Title: Cortical Excitability Assessment Using Paired Pulses
Acronym: PP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2014.865; 2014-A00495-42 (Other: ID-RCB)
Record Dates: First submitted 2014-09-09; First posted 2014-09-19 (Estimated); Last update posted 2019-10-23 (Actual); Status verified 2019-10

CONDITIONS: Focal Epilepsy
Keywords: pharmacoresistant focal epilepsy; cortical excitability; paired pulses; TMS; SEEG; DES
MeSH Terms: conditions — Epilepsies, Partial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- paired pulses cortical electrical stimulation (Experimental)
  Interventions: Other: paired pulses cortical electrical stimulation

INTERVENTIONS:
Other: paired pulses cortical electrical stimulation

SUMMARY:
The identification of the epileptogenic zone (EZ) during pharmacoresistant focal epilepsy presurgical assessment frequently requires intracranial recordings like stereo-electroencephalography (SEEG). Cortical direct electrical stimulation (DES) is commonly used during SEEG for functional mapping or to induce seizure.

However, the recording of seizures is sometimes insufficient to circumscribe the EZ and development of new biomarkers is necessary.

The cortex within the EZ is thought to be hyperexcitable. The "paired pulses" paradigm, using transcranial magnetic stimulation (TMS), allows determining the hemispheric cortical excitability level. The investigators hypothesize that paired pulses DES during SEEG could provide useful information for EZ identification.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years old
* Pharmacoresistant focal epilepsy patients undergoing a stereo-electroencephalographic recording
* Provide written consent to the study after receiving clear information
* Be a beneficiary or member of health insurance plan

Exclusion Criteria:

Patient with contraindication for MRI scanning

* Pregnancy
* Prohibition on participation in other research, apart from any other non-interventional research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-09-09 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Presence of a significant difference between the evoked responses to paired pulses cortical electrical stimulation of epileptogenic zone cortex and of normal cortex | between Day 7 and 21 (End of the stereoelectroencephalographic recordings)
  Low frequency single pulse electrical stimulation induces several cortico-cortical electroencephalographic responses: early-physiological and/or late-pathological. We expect different paired pulses modulation of those responses according the excitability level of the stimulated cortex (in terms of latency, amplitude, surface, frequency power)

SECONDARY OUTCOMES:
Presence of a difference of responses patterns between anatomic regions and/or lesion type | between Day 7 and 21 (End of the stereoelectroencephalographic recordings )
Presence of a difference between transcranial magnetic paired pulses stimulations and intracranial paired pulses cortical direct electrical stimulations | Between Day 7 and 21 (End of the stereoelectroencephalographic recordings)

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital neurologique de Lyon, Lyon, France